CLINICAL TRIAL: NCT00186511
Title: Expanding Rural Access: Distance Delivery of Support
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of California, Berkeley (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10AB-2801
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2006-12-05 (Estimated); Status verified 2006-12

CONDITIONS: Breast Cancer; Stress Disorders, Post-Traumatic; Depression
MeSH Terms: conditions — Breast Neoplasms; Stress Disorders, Post-Traumatic; Depression

INTERVENTIONS:
Behavioral: workbook/journal on coping with breast cancer
Behavioral: supportive expressive group therapy using videoconferencing

SUMMARY:
The major goal of this project is to test the feasibility and acceptability of using videoconferencing to provide support groups led by trained facilitators to rural women with breast cancer in northern California.

DETAILED DESCRIPTION:
Women with breast cancer in rural areas are likely exhaust their usual sources of psychosocial support while still facing challenges posed by breast cancer, but are unlikely to have access to professionally-led support groups. In this community-based project, we assessed the feasibility and acceptability of providing support groups to women with breast cancer in a large rural area using videoconferencing and a workbook journal, and we assessed the intervention's potential to reduce distress and increase emotional expression and self-efficacy for coping with cancer. Twenty-seven women in the Intermountain Region of northeastern California participated in 8-session support groups led by an oncology social worker by going to nearby videoconferencing sites. Feasibility and acceptability were demonstrated. Older as well as younger women were comfortable using videoconferencing and said the groups were valuable because they promoted information sharing and emotional bonds with other women with breast cancer. They emphasized the importance of a professional facilitator and identified advantages of using videoconferencing for support groups. Pretest and posttest comparisons showed significant decreases in depression and posttraumatic stress disorder symptoms. The results suggest that the intervention has the potential to provide a valuable service that is not readily available in rural communities.

ELIGIBILITY:
Inclusion Criteria:

* 1) has been diagnosed with breast cancer, and 2) is a woman

Exclusion Criteria:

* 1) under 21 years of age, and 2) does not speak and read English

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-11; Study Completion 2006-06

PRIMARY OUTCOMES:
Center for Epidemiological Studies Depression Scale
Posttraumatic Stress Checklist

SECONDARY OUTCOMES:
Cancer Behavior Inventory
Courtauld Emotional Control Scale

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Koopman, Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States